CLINICAL TRIAL: NCT06495203
Title: Establishing the Use of DARWEN AI Technology in Ophthalmology and Identifying Predictors of Treatment Intervals in nAMD and RVO
Brief Title: A Study to Understand the Usage of an Artificial Intelligence Technology Called DARWEN for Eye Disorders and to Find Out the Factors Influencing Treatment Frequencies in People With nAMD and RVO
Acronym: AIRSPEED
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22642
Record Dates: First submitted 2024-07-03; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Neovascular Age-related Macular Degeneration; Retinal Vein Occlusion
Keywords: nAMD; RVO; Central retinal vein occlusion; CRVO; Branch retinal vein occlusion; BRVO
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- nAMD patients, anti-VEGF naïve on treatment after July 2015: * Cluster A: Likely to require frequent injections
  * Cluster B: Probable to extend treatment interval
  * Cluster C: Likely to extend treatment interval
  Interventions: Drug: anti-VEGF treatment
- nAMD patients, anti-VEGF naïve on treatment before July 2015: * Cluster D: Likely to require frequent injections
  * Cluster E: Probable to extend treatment interval
  * Cluster F: Likely to extend treatment interval
  Interventions: Drug: anti-VEGF treatment
- nAMD patients, anti-VEGF experienced on treatment after July 2015: * Cluster G: Likely to require frequent injections
  * Cluster H: Likely to extend treatment interval
  Interventions: Drug: anti-VEGF treatment
- CRVO patients, anti-VEGF naïve on treatment after July 2015: * Cluster A: Likely to require continued anti-VEGF treatment
  * Cluster B: Likely to be off anti-VEGF treatment
  Interventions: Drug: anti-VEGF treatment
- BRVO patients, anti-VEGF naïve on treatment after March 2017: * Cluster C: Likely to require continued anti-VEGF treatment
  * Cluster D: Likely to be off anti-VEGF treatment
  Interventions: Drug: anti-VEGF treatment

INTERVENTIONS:
Drug: anti-VEGF treatment — Follow clinical practice/administration

SUMMARY:
This is an observational study in which data already collected from people with the eye disorders below are studied. In observational studies, only observations are made without participants receiving any advice or any changes to healthcare.

Neovascular age-related macular edema (nAMD): an eye disorder caused by the lack of oxygen in the retina. The lack of oxygen leads to the increase of a protein called vascular endothelial growth factor (VEGF). VEGF causes new, weak blood vessels to grow. These vessels can leak fluid or blood into the central part of the retina at the back of the eye (macula). This leads to blurring or a blind spot in the central (straight ahead) vision needed for reading or threading a needle.

Retinal vein occlusion (RVO): an eye disorder where a blood vessel that carries blood away from the retina (vein) becomes blocked. The blocked vein causes a lack of oxygen in the retina which leads to the increase of VEGF and then vision disturbances.

These eye disorders can be treated with a type of medicine called anti-vascular endothelial growth factor (anti-VEGF). Anti-VEGF treatment helps control the growth of new blood vessels in the eye and is given via injection into the eye.

DARWEN AI is a system using artificial intelligence (AI) technology. It has been proven that DARWEN AI can be used to extract data accurately and efficiently in multiple disease areas, including breast cancer, lung cancer, ambulatory care diseases and skin disorders.

The main purpose of this study is to validate if DARWEN AI can extract and sort through information from participants' health records accurately to identify those who need more frequent injections and those who do not.

The secondary purpose of this study is to use DARWEN AI to describe the factors influencing treatment frequencies in participants with nAMD or influencing treatment discontinuation in participants with RVO.

The data will come from the participants' information stored in EyeDoc Electronic Medical Records (EMR) at St. Joseph Health Care in London. Data collected are from January 1, 2009, to May 31, 2023.

ELIGIBILITY:
Inclusion Criteria:

* All patients with the diagnosis of nAMD or RVO (Branch or Central) who are patients of Dr. Tom Sheidow listed in the EyeDoc EHR with available patient records from Jan 1, 2009 to May 31, 2023.

Exclusion Criteria:

* Not applicable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with the diagnosis of nAMD or RVO (Branch or Central) who are patients of Dr. Tom Sheidow listed in the EyeDoc Electronic Health Record (EHR) with available patient records from Jan 1, 2009 to May 31, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 1350 (Actual)
Dates: Start 2023-11-02 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Validation of DARWEN™ AI. | Retrospective data analysis from January 1, 2009 to May 31, 2023.
  Based on defined objective clinical eligibility criteria, the EMR data set was divided into four cohorts using Pentavere's proprietary AI engine DARWEN™. The following ophthalmology-specific variables were validated against a manual review: diagnosis of nAMD, diagnosis of RVO including CRVO and BRVO, treatment intervals of anti-VEGF treatment grouped as < Q8 weeks or ≥ Q8 weeks for nAMD patients, discontinuation of anti-VEGF treatment for RVO patients, and the final outputted cohorts. The manual review was performed on a random selection of 25 patients from each of the four cohorts (100 patients total). Two trained manual abstractors classified these patients according to the rules outlined in the objective cohort criteria. They aligned on a consensus for each patient and compared with the DARWEN™cohorts. Pentavere then provided a success rate for the accuracy of the classification.

SECONDARY OUTCOMES:
Summary of baseline demographics reported as number of participants with different categories. | Retrospective data analysis from January 1, 2009 to May 31, 2023.
  Age, sex.
Summary of clinical characteristics reported as number of participants with different categories. | Retrospective data analysis from January 1, 2009 to May 31, 2023.
  Baseline ophthalmology characteristics, ocular comorbidities, other comorbidities, family history, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Bayer, Mississauga, Canada

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.